CLINICAL TRIAL: NCT05469477
Title: Behavioral Interventions to Increase Seat Belt Wearing and Decrease Handheld Phone Use While Driving
Brief Title: Increasing Seat Belt Wearing and Decreasing Handheld Phone Use While Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: General Motors (GM) (Unknown)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 851411
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Distracted Driving; Impaired Driving; Driving Behaviors
Keywords: Habit Formation; Financial Incentives; Phone Use While Driving; Seat Belt Wearing
MeSH Terms: interventions — NEUROG1 protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Other): Participants are asked to buckle up and not engage in handheld phone use while driving. No further messaging will be provided about their behavior, and participants will not receive financial incentives for avoiding risky driving behavior.
  Interventions: Behavioral: Weekly SMS Support text
- Behavioral Engagement (Experimental): Participants will receive a multicomponent safer driving intervention based on behavioral science. This will include persuasive education, WOOP (mental contrasting with implementation intentions) and customized habit tips.
  Interventions: Behavioral: Persuasive education; Behavioral: WOOP (aka, mental contrasting with implementation intentions., Wish, Outcome, Obstacle, Plan); Behavioral: Customized Habit Tips; Behavioral: Weekly SMS Support text; Behavioral: Weekly SMS Encouragement
- Raffle incentive + behavioral engagement (Experimental): Participants will receive the entire multicomponent safer driving behavioral intervention from arm 2. Participants will also be eligible for the Raffle Financial incentive, where participants can earn prize money for seat belt adherence and/or no phone use while driving.
  Interventions: Behavioral: Persuasive education; Behavioral: WOOP (aka, mental contrasting with implementation intentions., Wish, Outcome, Obstacle, Plan); Behavioral: Customized Habit Tips; Behavioral: Raffle Financial Incentive; Behavioral: Weekly SMS Support text; Behavioral: Weekly SMS Encouragement
- Shared pot incentive + behavioral engagement (Experimental): Participants will receive the entire multicomponent safer driving behavioral intervention from arm 2. This arm will be identical to Arm 3, except there will be a shared pot financial incentive instead of a raffle. Participants that abstain from phone use while driving and seat belt adherence earn an equal share of prize money allocated for the entire group.
  Interventions: Behavioral: Persuasive education; Behavioral: WOOP (aka, mental contrasting with implementation intentions., Wish, Outcome, Obstacle, Plan); Behavioral: Customized Habit Tips; Behavioral: Shared Pot Financial Incentive; Behavioral: Weekly SMS Support text; Behavioral: Weekly SMS Encouragement

INTERVENTIONS:
Behavioral: Persuasive education — The research team will use psychology and communications research to present information about seat belts and distracted driving in a way that builds intrinsic motivation to change. Because positively framed messages are more effective at promoting seat belt wearing, the team's messaging will employ this framing. Education will address common reasons that survey participants give for not consistently buckling up or for phone use while driving.
  Arms: Behavioral Engagement; Raffle incentive + behavioral engagement; Shared pot incentive + behavioral engagement
Behavioral: WOOP (aka, mental contrasting with implementation intentions., Wish, Outcome, Obstacle, Plan) — Participants will receive an intervention on improving driving behavior with a specific goal in mind and how to reach that goal. Participants will do this by thinking through 4 parts: a wish, an outcome, an obstacle and a plan. This has been shown to build motivation, and help achieve the desired change.
  Arms: Behavioral Engagement; Raffle incentive + behavioral engagement; Shared pot incentive + behavioral engagement
Behavioral: Customized Habit Tips — Participants will receive weekly text-message tips, informed by findings from survey responses, plus reminders to address stated obstacles.
  Arms: Behavioral Engagement; Raffle incentive + behavioral engagement; Shared pot incentive + behavioral engagement
Behavioral: Raffle Financial Incentive — Each week, participants who adhere to seat belt use or abstain from phone use while driving get a chance at prize money. One winner will be randomly chosen for each target behavior and earn prize money; the rest will not receive compensation.
  Arms: Raffle incentive + behavioral engagement
Behavioral: Shared Pot Financial Incentive — This will be identical to the raffle incentive, except that each week participants who adhere to seat belt use or abstain from phone use while driving will be guaranteed an equal share of prize money.
  Arms: Shared pot incentive + behavioral engagement
Behavioral: Weekly SMS Support text — Participants will receive a support SMS to troubleshoot, etc. if the Way to Drive app is not collecting trip data.
Behavioral: Weekly SMS Encouragement — Those who have a perfect streak going midway through each week will receive an additional encouraging message cheering them on.
  Arms: Behavioral Engagement; Raffle incentive + behavioral engagement; Shared pot incentive + behavioral engagement

SUMMARY:
The study team is proposing to conduct a randomized controlled trial to determine the effectiveness of behavioral and financial incentives on phone use while driving and seat belt adherence. Each arm will receive a support text if their app is not collecting data. The behavioral engagement intervention includes persuasive education, mental contrasting with implementation intentions, customized habit tips, weekly feedback about participants' streaks, and encouraging SMS texts. The two financial incentive interventions add on weekly raffles or shared pots for participants with perfect streaks.

ELIGIBILITY:
Inclusion Criteria:

* Are a GM/OnStar customer.
* Are 18 or older.
* Meet minimum trip requirements.
* Uses vehicle with OnStar
* At least 5 weeks of baseline trip data with >=8 trips/week at baseline on average
* Baseline seat belt use <= 75% on trips less than 2 miles and <= 90 on trips greater than 2 miles
* English reading ability
* Have an email address
* Have a smartphone with iPhone iOS 12 or later or Android OS 7 or later

Exclusion Criteria:

* You are unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Proportion of trips with seat belt use | 105 days
  Calculated as the number of trips during which a driver's seat belt click was detected, divided by total number of trips (defined as 1/10 of a mile or greater).

SECONDARY OUTCOMES:
Seconds of active (handheld) phone use per hour of driving | 105 days
  This is a composite outcome that measures the proportion of total trip time in which the driver is engaged in handheld phone call use or non-call handheld use (e.g. texting, swiping, and typing), as measured by the Way to Drive app.

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Delgado, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dingus TA, Guo F, Lee S, Antin JF, Perez M, Buchanan-King M, Hankey J. Driver crash risk factors and prevalence evaluation using naturalistic driving data. Proc Natl Acad Sci U S A. 2016 Mar 8;113(10):2636-41. doi: 10.1073/pnas.1513271113. Epub 2016 Feb 22. PMID 26903657
- [Background] Gershon P, Sita KR, Zhu C, Ehsani JP, Klauer SG, Dingus TA, Simons-Morton BG. Distracted Driving, Visual Inattention, and Crash Risk Among Teenage Drivers. Am J Prev Med. 2019 Apr;56(4):494-500. doi: 10.1016/j.amepre.2018.11.024. Epub 2019 Feb 21. PMID 30799162
- [Background] Klauer SG, Guo F, Simons-Morton BG, Ouimet MC, Lee SE, Dingus TA. Distracted driving and risk of road crashes among novice and experienced drivers. N Engl J Med. 2014 Jan 2;370(1):54-9. doi: 10.1056/NEJMsa1204142. PMID 24382065
- [Background] Simons-Morton BG, Guo F, Klauer SG, Ehsani JP, Pradhan AK. Keep your eyes on the road: young driver crash risk increases according to duration of distraction. J Adolesc Health. 2014 May;54(5 Suppl):S61-7. doi: 10.1016/j.jadohealth.2013.11.021. PMID 24759443
- [Derived] Ebert JP, Yan R, Friday S, Small D, McDonald CC, Bartolozzi K, Delgado MK. Behavioral Interventions for Increasing Seat Belt Use and Decreasing Distracted Driving Using Telematics: A National Randomized Trial. Am J Public Health. 2025 May;115(5):758-768. doi: 10.2105/AJPH.2024.307980. Epub 2025 Mar 13. PMID 40080744